CLINICAL TRIAL: NCT04997304
Title: Utilizing Advances in Digital Inhaler Technology to Understand Heterogeneous Treatment Responses to Biologics in Severe Asthma
Brief Title: Teva Asthma Predictive Analytics Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Principal Investigator, Njira Lugogo, Associate Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00189756
Record Dates: First submitted 2021-07-11; First posted 2021-08-09 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Asthma
Keywords: Adults; Severe persistent; AirDuo Digihaler; ProAir Digihaler
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AirDuo and ProAir (Experimental): This trial includes using the inhaler (AirDuo®) Digihaler™ and rescue inhalers (ProAir®) Digihaler™.
  Interventions: Combination Product: AirDuo Digihaler; Combination Product: ProAir Digihaler

INTERVENTIONS:
Combination Product: AirDuo Digihaler — Participants will receive the AirDuo® Digihaler™ at a dose that is equivalent to the participants' current inhaled therapy dose. Most participants will likely require the high dose inhaler: 232/14 device. This medication will be administered twice daily. The study and treatment will last 1 year.
  Participants will also use a home spirometry device and smart device application (app) will be used to track medication usage and allow users to self-assess their respiratory symptoms on a daily basis.
Combination Product: ProAir Digihaler — Participants will receive the ProAir® Digihaler™ 90mcg at a dose that is equivalent to the participants' current inhaled therapy dose. Most participants will likely require the high dose inhaler: 232/14 device. The ProAir® Digihaler™ will be utilized up to six times per day as needed for acute asthma symptoms. The study and treatment will last 1 year.

SUMMARY:
This trial is being completed to determine baseline inhalation parameters and patterns of use in patients receiving treatment with TEVA digital inhalers, to develop predictive models for asthma exacerbations and response to biologics using data collected from these devices.

Enrolled participants will complete questionnaires along with other study specific procedures. Additionally, in-person and phone visits will be performed.

DETAILED DESCRIPTION:
All participants were provided an AirDuo® Digihaler™ and ProAirDuo® Digihaler™, which the participants could choose to use or not. This trial did not restrict participants from using other asthma treatments in addition to or in lieu of the Digihalers.

ELIGIBILITY:
Inclusion Criteria:

* A history of severe persistent asthma as defined by European Respiratory Society (ERS) and American Thoracic Society (ERS/ATS) criteria which includes the presence of poor asthma control on high dose inhaled corticosteroid (ICS) and a long-acting beta-agonist (CS/LABA) or the need for high dose ICS/LABA to maintain asthma control or oral steroids for maintenance therapy for more than 50% of the prior year.
* Presence of current biologic use or planned initiation of biologics following study enrollment
* Patients will be categorized on the basis of asthma control (Asthma Control Test (ACT)< 19 will be considered poor asthma control). The study will cap the patients with good asthma control at 30% and will no longer enroll those patients once the strata have been fully enrolled.
* Willingness to switch maintenance inhalers to AirDuo® Digihaler™ and to use ProAir® Digihaler™ for rescue therapy. Use of nebulized albuterol will be discouraged but not prohibited.
* Can read and communicate in English and is familiar with and is willing to use his/her own smart device and download and use the study application
* Ability to provide informed consent.
* The patient must be willing and able to comply with study requirements and restrictions

Exclusion Criteria:

* Clinically important pulmonary disease other than asthma including Chronic obstructive pulmonary disease (COPD), bronchiectasis, pulmonary fibrosis, cystic fibrosis, or other lung disease
* Any disorder that is either not stable or could in the opinion of the investigator affect the ability of the subject to safely participate in the study or could adversely affect study results.
* History of human immunodeficiency virus or other immunodeficiency syndrome
* Malignancy other than skin cancer that has occurred within the past year and that will impact survival thus limit participation in the clinical trial
* History of chronic alcohol abuse or drug use
* Any life-threatening diseases that will impact the patient's ability to complete the 12-month study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Njira Lugogo, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AirDuo and ProAir: This trial includes using the inhaler (AirDuo®) Digihaler™ and rescue inhalers (ProAir®) Digihaler™.
  AirDuo Digihaler: Participants will receive the AirDuo® Digihaler™ at a dose that is equivalent to the participants' current inhaled therapy dose. Most participants will likely require the high dose inhaler: 232/14 device. This medication will be administered twice daily. The study and treatment will last 1 year.
  Participants will also use a home spirometry device and smart device application (app) will be used to track medication usage and allow users to self-assess their respiratory symptoms on a daily basis.
  ProAir Digihaler: Participants will receive the ProAir® Digihaler™ 90mcg at a dose that is equivalent to the participants' current inhaled therapy dose. Most participants will likely require the high dose inhaler: 232/14 device. The ProAir® Digihaler™ will be utilized up to six times per day as needed for acute asthma symptoms. The study and treatment will last 1 year.
Period: Overall Study
Arm/Group | AirDuo and ProAir
Started | 100
Completed | 74
Not Completed | 26
Not completed — Lost to Follow-up | 11
Not completed — Death | 1
Not completed — Withdrawal by Subject | 14

BASELINE CHARACTERISTICS:
Arm/Group | AirDuo and ProAir
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 94
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 16
  White | 76
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Daily Doses of ProAir® Digihaler™
Description: This outcome measured participant adherence to using the ProAir® Digihaler™. All participants were provided the Digihaler device, which they could choose to use or not. Subject-specific result was calculated as the sum total of doses taken by participant divided by their number of days of follow-up.
Time Frame: up to 1 year
Population: Because the outcome measure concerned adherence, all participants were included in this outcome, regardless of whether they chose to use the ProAir® Digihaler™.
Measure: Mean (Standard Deviation); unit: doses per day
Groups:
- ProAir® Digihaler: Participants were provided with the ProAir® Digihaler™ 90mcg inhaler, which they could choose to use or not. If taken, participants would receive a dose that was equivalent to the participants' current inhaled therapy dose. The ProAir® Digihaler™ will be utilized up to six times per day as needed for acute asthma symptoms. The study and treatment will last 1 year.
  Participants will also use a home spirometry device and smart device application (app) will be used to track medication usage and allow users to self-assess their respiratory symptoms on a daily basis.
Arm/Group | ProAir® Digihaler
Number analyzed (Participants) | 100
doses per day | 0.55 (0.95)

2. Primary Outcome: Mean Number of Daily Doses AirDuo® Digihaler™.
Description: This outcome measured participant adherence to using the AirDuo® Digihaler™. All participants were provided the Digihaler, which they could choose to use or not. Subject-specific result was calculated as the sum total of doses for a given participant divided by their number of days of follow-up.
Time Frame: up to 1 year
Population: Because the outcome measure concerned adherence, all participants were included in this outcome, regardless of whether they chose to use the AirDuo® Digihaler™.
Measure: Mean (Standard Deviation); unit: doses per day
Groups:
- AirDuo® Digihaler: Participants were provided with the AirDuo® Digihaler™ inhaler, which they could choose to use or not. If taken, participants will receive the AirDuo® Digihaler™ at a dose that is equivalent to the participants' current inhaled maintenance therapy dose. Most participants will likely require the high dose inhaler: 232/14 device. This medication will be administered twice daily. The study and treatment will last 1 year.
  Participants will also use a home spirometry device and smart device application (app) will be used to track medication usage and allow users to self-assess their respiratory symptoms on a daily basis.
Arm/Group | AirDuo® Digihaler
Number analyzed (Participants) | 100
doses per day | 0.99 (0.76)

3. Primary Outcome: Median Number of Daily Doses of ProAir® Digihaler™
Description: This outcome measured participant adherence to using the ProAir® Digihaler™. All participants were provided the Digihaler, which they could choose to use or not. Subject-specific result was calculated as the 50th percentile value of all daily dose totals (or the average of two 50th percentile values if there was a tie) calculated over the number of days of follow-up.
Time Frame: up to 1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: doses per day
Arm/Group | ProAir® Digihaler
Number analyzed (Participants) | 100
doses per day | 0.21 [0.03 to 0.52]

4. Primary Outcome: Median Number of Daily Doses of AirDuo® Digihaler™
Description: This outcome measured participant adherence to using the AirDuo® Digihaler™. All participants were provided the Digihaler, which they could choose to use or not. Subject-specific result was calculated as the 50th percentile value of all daily dose totals (or the average of two 50th percentile values if there was a tie) calculated over the number of days of follow-up.
Time Frame: up to 1 year
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: doses per day
Arm/Group | AirDuo® Digihaler
Number analyzed (Participants) | 100
doses per day | 0.99 [0.21 to 1.66]

5. Secondary Outcome: Maintenace Inhaler Adherence Rates
Description: This outcome measured participant adherence to using the AirDuo® Digihaler™. All participants were provided the Digihaler, which they could choose to use or not. Adherence rates were measured by the following: High (>80% of puffs), moderate (50-80% of puffs), and low levels (<50% of puffs) of adherence to maintenance inhalers over the course of the trial.
Time Frame: up to 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | AirDuo® Digihaler
Number analyzed (Participants) | 100
Participants
  High (>80% of puffs) | 23
  Moderate (50-80% of puffs) | 25
  Low levels (<50% of puffs) | 52

6. Secondary Outcome: Participants Who Achieved Non-response, Partial Response, and Complete Response to Biologics
Description: All participants were provided the AirDuo® and ProAir® Digihalers, which they could choose to use or not. Responses were categorized as non-response, partial response, and complete response on the basis of five factors: a 50% reduction in exacerbations, any reduction in maintenance oral corticosteroids (OCS) dose, change of at least 10% in forced expiratory volume in one second (FEV1), improvement of 3 points in asthma control test (ACT) score, and patient perception of global improvement in asthma. Non-response indicated that a participant had no response to any of the 5 factors. Partial response indicated that a participant responded to at least 1 factor. Complete response indicated that a participant responded to all 5 factors.
Time Frame: up to 1 year
Population: Because the outcome measure concerned response to biologics, all participants were included in this outcome, regardless of whether they chose to use either Digihaler or not.
Measure: Count of Participants; unit: Participants
Arm/Group | AirDuo and ProAir
Number analyzed (Participants) | 100
Participants
  Non-response | 3
  Partial response | 82
  Complete response | 15

7. Secondary Outcome: Change in Mean Peak Inhalation Volume
Description: Peak inhalation volume is the maximum air volume a person can breathe in during a deep inhalation, serving as an indicator of lung capacity and respiratory function. Peak inhalation volume was measured by the digital inhaler at the end of inhalation. This measures the maximum volume that the participant was able to draw into their lungs. Larger numbers indicated healthier lungs.
Time Frame: baseline to 1 year
Population: Measurements were taken for those participants who experienced an exacerbation and compared to their baseline values. Because the ProAir is a rescue inhaler, not all individuals used it, so the number of participants involved is smaller.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | AirDuo and ProAir
Number analyzed (Participants) | 48
milliliters
  Baseline - AirDuo | 2436.48 (1328.27)
  Follow Up/Exacerbation - AirDuo | 2041.79 (803.00)
  Baseline - ProAir: number analyzed (Participants) | 44
  Baseline - ProAir | 2147.69 (1201.34)
  Follow Up/Exacerbation - ProAir: number analyzed (Participants) | 44
  Follow Up/Exacerbation - ProAir | 1833.74 (806.61)
Statistical Analysis 1: Comparison: AirDuo and ProAir; This analysis applies only to comparison of baseline and exacerbation for AirDuo; Test type: Other — Test of paired differences; p = 0.0019, t-test, 2 sided; Paired t-test
Statistical Analysis 2: Comparison: AirDuo and ProAir; This analysis applies only to comparison of baseline and exacerbation for ProAir; Test type: Other — Test of paired differences; p = 0.0020, t-test, 2 sided; Paired t-test

8. Secondary Outcome: Change in Mean Inspiratory Time
Description: Inspiratory time was the total time taken to complete an inspiration (i.e., breathing in). Results were differences between the baseline and exacerbation measurements.
Time Frame: baseline to 1 year
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | AirDuo and ProAir
Number analyzed (Participants) | 48
Seconds
  Baseline - AirDuo | 2002.99 (853.03)
  Follow Up/Exacerbation - AirDuo | 1755.44 (692.41)
  Baseline - ProAir: number analyzed (Participants) | 44
  Baseline - ProAir | 2268.19 (919.78)
  Follow Up/Exacerbation - ProAir: number analyzed (Participants) | 44
  Follow Up/Exacerbation - ProAir | 1982.48 (756.34)
Statistical Analysis 1: Comparison: AirDuo and ProAir; This analysis applies only to comparison of baseline and exacerbation for AirDuo; Test type: Other — Test of paired differences; p = 0.0008, t-test, 2 sided; Paired t-test
Statistical Analysis 2: Comparison: AirDuo and ProAir; This analysis applies only to comparison of baseline and exacerbation for ProAir; Test type: Other — Test of paired differences; p = 0.0003, t-test, 2 sided; Paired t-test

9. Secondary Outcome: Change in Mean Peak Inspiratory Flow (PIF)
Description: PIF is the maximum rate of airflow a person can inhale using an inhaler after a full breath. PIF was measured by the ProAir® Digihaler™ and AirDuo® Digihaler™. Results indicate the changes between the baseline and exacerbation measurements.
Time Frame: baseline up to 1 year
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liters per minute
Arm/Group | AirDuo and ProAir
Number analyzed (Participants) | 48
Liters per minute
  Baseline - AirDuo | 103.41 (35.02)
  Follow Up/Exacerbation - AirDuo | 99.04 (29.58)
  Baseline - ProAir: number analyzed (Participants) | 44
  Baseline - ProAir | 79.60 (27.08)
  Follow Up/Exacerbation - ProAir: number analyzed (Participants) | 44
  Follow Up/Exacerbation - ProAir | 77.14 (23.61)
Statistical Analysis 1: Comparison: AirDuo and ProAir; This analysis applies only to comparison of baseline and exacerbation for AirDuo; Test type: Other — Test of paired differences; p = 0.04, t-test, 2 sided; Paired t-test
Statistical Analysis 2: Comparison: AirDuo and ProAir; This analysis applies only to comparison of baseline and exacerbation for ProAir; Test type: Other — Test of paired differences; p = 0.0965, t-test, 2 sided; Paired t-test

10. Secondary Outcome: Change in Mean Forced Expiratory Volume in One Second (FEV1)
Description: FEV1 was measured using the Go Spiro Spirometer. Results indicate the difference between the baseline and exacerbation measurements.
Time Frame: baseline up to 1 year
Population: Measurements were taken for those participants who experienced an exacerbation and compared to their baseline values. Home spirometry was not consistently used by all participants.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | AirDuo and ProAir
Number analyzed (Participants) | 20
Liters
  Baseline | 66.07 (20.34)
  Follow Up/Exacerbation | 68.43 (19.47)

11. Other Pre Specified Outcome: Number of Exacerbations
Time Frame: up to 1 year
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Number of Hospitalizations
Time Frame: up to 1 year
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Number of Emergency Room Visits
Time Frame: up to 1 year
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Mean Asthma Control Test (ACT) Score
Time Frame: up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: Adverse event data in arms 2, 3, and 4 reflect instances where an adverse event occurred within 1 month of the participant using the named intervention. Data reflects only participant use of the AirDuo and ProAir. Note: some participants on their own accord used a different product instead of, or in conjunction with, the AirDuo or ProAir. Usage of these other products, not being part of this pragmatic trial, were not tracked.
Groups:
- Not Using Either AirDuo or ProAir: Participants used neither inhaler during the course of the trial.
- After Using AirDuo: Data reflects participants who experienced an AE within 1 month of using the AirDuo.
- After Using ProAir: Data reflects participants who experienced an AE within 1 month of using the ProAir. 73 participants used ProAir at all during the trial.
- After Using Both AirDuo and ProAir: Data reflects participants who experienced an AE within 1 month of using both AirDuo and ProAir inhalers together.73 participants used both AirDuo and ProAir during the trial.
Arm/Group | Not Using Either AirDuo or ProAir | After Using AirDuo | After Using ProAir | After Using Both AirDuo and ProAir
All-Cause Mortality (participants affected / at risk) | 1/16 | 0/84 | 0/73 | 0/73
Serious Adverse Events (participants affected / at risk) | 5/16 | 0/84 | 2/73 | 8/73
Other Adverse Events (participants affected / at risk) | 7/16 | 7/84 | 1/73 | 18/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Not Using Either AirDuo or ProAir (N=16) | After Using AirDuo (N=84) | After Using ProAir (N=73) | After Using Both AirDuo and ProAir (N=73)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Tremors & Generalized Weakness (General disorders) | 0 | 0 | 0 | 1
Influenza A (Infections and infestations) | 0 | 0 | 0 | 1
Covid 19 (Infections and infestations) | 0 | 0 | 1 | 0
Adrenal Crisis (Endocrine disorders) | 1 | 0 | 0 | 0
Gastroparesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Graham Negative Rod Bacteremia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Post-surgical low oxygen (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Not Using Either AirDuo or ProAir (N=16) | After Using AirDuo (N=84) | After Using ProAir (N=73) | After Using Both AirDuo and ProAir (N=73)
Covid 19 (Infections and infestations) | 2 | 4 | 1 | 9
Sinus Infection (Infections and infestations) | 1 | 1 | 0 | 5
Upper Respiratory Infection (Infections and infestations) | 4 | 2 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT04997304/Prot_SAP_000.pdf